CLINICAL TRIAL: NCT06565130
Title: Attention Skills of Wheelchair Basketball Players: Occupational Therapy Intervention
Brief Title: Wheelchair Basketball and Attention Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Sultan Akel, Lecturer, Bezmialem Vakif University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022/286
Record Dates: First submitted 2023-07-24; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Physical Disability
Keywords: attention skills; occupational therapy; wheelchair basketball

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Attention Skills Training (Other): Intervention plan, which will begin by talking about the importance of attention in sports; It will consist of different tasks that include sub-parameters of attention, such as maintaining attention, shifting attention, focusing attention and splitting attention.
  Interventions: Other: Attention skills training

INTERVENTIONS:
Other: Attention skills training — Attention skills program planned with occupational therapy principles

SUMMARY:
The goal of this interventional study is to evaluate the effect of attention training on performance in wheelchair basketball players. The main question it aims to answer is:

Does attention training have an effect on the performance of wheelchair basketball players? Participants will participate attention training from an occupational therapy perspective.

DETAILED DESCRIPTION:
The attention skills of the athletes will be evaluated with a competition-like designed assessment session. Then, the planned 10-week intervention program will be carried out as one session per week. After the intervention program, the evaluation session will be repeated and the results will be recorded. Then, it will be evaluated whether there is improvement in the attention skills of the athletes. The results obtained will be important for athletes, coaches and professionals working in this field.

ELIGIBILITY:
Inclusion Criteria:

* Actively active in a regional wheelchair basketball team for at least 6 months.
* Volunteering to participate in the research.
* Being literate.

Exclusion Criteria:

* Having a neurological or cognitive disorder other than a physical disability.
* Being colorblind.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2023-03-12 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
The number of successful shots | 10 week
  The number of mistakes made during the physical activity and track will be recorded as one.Athletes can make mistakes at any stage of the course (depending on their attention skills). Each mistake will be considered a numerical unit and will be written as one piece.

SECONDARY OUTCOMES:
The time to complete the track and each stage | 10 week
  The time spent by athletes on each stage of the track and the time it takes to complete the physical activity will be recorded. These times will be considered as a outcome measures.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No